CLINICAL TRIAL: NCT03370549
Title: Developing an Intervention to Promote API Women's Sexual and Mental Health
Brief Title: Asian Women's Action in Resilience and Empowerment
Acronym: AWARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: Rutgers University (Other)
Responsible Party: Principal Investigator, Hyeouk Hahm, Associate Professor, Boston University Charles River Campus
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: BostonUCRC
Record Dates: First submitted 2017-11-29; First posted 2017-12-12 (Actual); Last update posted 2017-12-12 (Actual); Status verified 2017-12

CONDITIONS: Mental Health Disorder
Keywords: Mental health; Suicide; Sexual risk behaviors
MeSH Terms: conditions — Mental Disorders; Psychological Well-Being; Suicide

STUDY DESIGN:
Intervention Model Description: We employed a two-arm randomized clinical trial to test the preliminary feasibility, safety, and efficacy for AWARE intervention comparing the AWARE intervention group (n=48) with the wait-list group (n =48).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AWARE intervention (Experimental): Group psychotherapy intervention for Asian-American women
  Interventions: Behavioral: AWARE intervention
- Waitlist control (Other): Delayed AWARE intervention for Asian-American women
  Interventions: Behavioral: AWARE intervention

INTERVENTIONS:
Behavioral: AWARE intervention — Group psychotherapy for Asian-American women

SUMMARY:
Our objective for this R34 is to develop gender/culture specific and trauma informed group psychotherapy intervention designed to treat Chinese-, Korean-, and Vietnamese-American young women with histories of interpersonal violence trauma. The intervention is called Asian Women's Action for Resilience and Empowerment (AWARE).

DETAILED DESCRIPTION:
Recent epidemiological studies document two emerging public health problems among Asian-Pacific Islander (API) women in the US:

1. A growing incidence of HIV/AIDS. Although the prevalence of HIV/AIDS among APIs is low compared to those among Blacks, Whites, and Hispanics, HIV infection among APIs significantly increased (44%) between 2004 and 2007. Additionally, 75% of HIV transmission among API women is through heterosexual intercourse, which is substantially higher than percentages among other racial/ethnic groups of women.
2. Poor mental health functioning exhibited by completed suicide rates. Young API women (ages 15 to 34) have not only the highest rates of completed suicide compared to other women of the same age in the US, but also experienced the largest growth in rates of suicide over the past decade.

Our preliminary studies using both quantitative and qualitative methods found strong links between past trauma and poor sexual and mental health outcomes. For API women, reporting a history of forced sex was associated with higher odds of severe depression, substance use, getting pregnant, and HIV risk behaviors compared to API women who did not report a history of forced sex. API women continue to be vulnerable given their lower rates of HIV testing, lower mental health utilization, and premature dropout rates in mental health treatment compared to other racial groups. So far, no existing intervention targets both sexual health and mental health problems among API women. Specifically, this study builds upon data on API women from prior NIMH-funded work as the foundation for our intervention.

ELIGIBILITY:
Inclusion Criteria:

* self-identify as female;
* are unmarried;
* are between the ages 18 and 35;
* are of Chinese, Korean, and/or Vietnamese descent;
* are 1.5 (immigrated to the US before the age of 18) or 2nd (US-born children of 1st generation immigrants) generation;
* are fluent in English;
* have a mobile phone with text messaging;
* have had penile-vaginal intercourse in their lifetime;
* have a history of exposure to at least one of five selected criteria in the Traumatic Life Events Questionnaire (TLEQ). These criteria include: beaten by stranger, death threat, childhood physical abuse, family violence, and partner physical assault;

Exclusion Criteria:

* at current significant risk of homicidal or suicidal behavior
* having symptoms of psychosis;
* have previously experienced natural disasters or other non-violent trauma;
* are of mixed race other than Korean-, Chinese-, or Vietnamese-Americans;

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 96 (Actual)
Dates: Start 2013-08-01 (Actual); Primary Completion 2016-06-23 (Actual); Study Completion 2017-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Sexual Risk Behaviors | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  AIDS Risk Behavior Assessment (ARBA) was used. Sexual risk behaviors were defined as engaging in unprotected sex, having multiple sex partners, and engaging in anal sex. Engagement in unprotected sex was assessed by asking participants, "Of those times that you had vaginal sex in the past three months, how often did you or your partner use condoms/latex protection?'' Responses were scored 0 for "never used a condom," "some of the time," "half of the time," "more than half of the time" and 1 for "every time." Having multiple sex partners was assessed by the question: "How many female/male sex partners have you had in the past three months?" Responses were coded dichotomously as 0 for none or one sexual partner and 1 for more than one sexual partner. Engagement in anal sex was assessed by the question, "How many times in the past three months did you have anal sex?" Responses were dichotomized as 0 for none, and 1 for one or more times.

SECONDARY OUTCOMES:
Change in Depressive Symptoms | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The Center for Epidemiological Studies Depression Scale (CES-D) is a 20-item self-report questionnaire designed to assess depressive symptomatology. For each item, participants reported their status over the past two weeks using a Likert-type scale ranging from rarely or never (0) to most days or always (3). Responses were summed to create a total symptom score ranging from 0 to 60. The CES-D has demonstrated very high internal consistency, reliability and validity. The internal consistency of our sample ranged from .86 to .92.
Change in Substance Use | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  Addiction Severity Index (ASI) is a self-report questionnaire for patients who present for substance abuse treatment. The instrument gathers information about seven areas of a patients life: medical, employment/support, drug and alcohol use, legal, family history, family/social relationships. The scale has Cronbach's alpha of alcohol section of 0.75 and for Drug section is 0.70. This measure was used in testing SS for women who suffered from substance use and PTSD.
Change in Mental Distress | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The General Mental Distress Index (GMDI) is a 21-item scale screening for symptoms of depression, anxiety, suicidal ideation, and other aspects of mental and emotional distress. Each item is scored 1 for "yes" and 0 for "no." A score of 4-6 indicates clinically-significant symptoms, and a score of 7+ indicates acute distress with the possibility of reoccurring mental health problems.

OTHER OUTCOMES:
Change in PTSD Symptoms | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The PTSD Checklist, Civilian version (PCL-C) is a 17-item self-report measure of PTSD symptom severity. Each item corresponds to a PTSD symptom outlined in the fourth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-IV). Participants reported both the frequency and intensity of their experiences of PTSD symptoms over the past three months on a 5-point scale ranging from low to high. Symptom severity was computed by summing the frequency and intensity scores. Total scores ranged from 17 to 85, with a score of 50 used as the cutoff to assess a diagnosis of PTSD.
Change in Safety Outcome | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The Columbia-Suicide Severity Rating Scale (C-SSRS) was used to assess history of suicidal ideation and suicidal intent. Participants who reported yes to either one of the following questions were classified as having suicidal ideation--wished to be dead, thought of killing yourself, and thought about how to do this. Suicidal intent was measured with answering yes to either one of having intention of acting on thoughts of killing yourself as well as having worked out the details of how to do it. At baseline (T0), lifetime suicidal outcomes were measured and. For the post intervention evaluations (T1, T2), suicidal outcomes of the past 30 days were measured.
Change in HIV Knowledge | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The HIV-Knowledge Questionnaire (HIV-KQ) is a 45-item assessment on knowledge pertaining to HIV. Statements are responded to in a true/false/don't know format, addressing topics of prevention (i.e. safe sex practices), transmission (i.e. sexual transmission and other modes) and consequences (i.e. testing and treatment). The HIV-KQ exhibits a high internal consistency, with Cronbach's alpha = 0.91.
Change in Self-Efficacy Scale | Outcomes will be measured at: baseline, up to 12 weeks after the baseline, 3 months post intervention
  The Self-efficacy Scale for Limiting HIV Risk Behaviors (LHRB) contains 9 statements on self-efficacy pertaining to HIV risk behaviors. Participants are asked to rate how sure they are that they could perform each statement (0= not sure at all to 4=very sure).
Feasibility Outcome | 8 weeks of treatment
  Participant retention was evaluated using the number of sessions attended. The "completers" of the intervention were defined as those who attended at least 80% of the sessions. Similar definitions have been used in other studies.

CONTACTS AND LOCATIONS:
Overall Officials: Hyeouk Hahm, Ph.D., LCSW, Principal Investigator — Boston University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hahm HC, Lee J, Rough K, Strathdee SA. Gender power control, sexual experiences, safer sex practices, and potential HIV risk behaviors among young Asian-American women. AIDS Behav. 2012 Jan;16(1):179-88. doi: 10.1007/s10461-011-9885-2. PMID 21259042
- [Background] Hahm HC, Kolaczyk E, Lee Y, Jang J, Ng L. Do Asian-American women who were maltreated as children have a higher likelihood for HIV risk behaviors and adverse mental health outcomes? Womens Health Issues. 2012 Jan-Feb;22(1):e35-43. doi: 10.1016/j.whi.2011.07.003. Epub 2011 Aug 26. PMID 21872488
- [Background] Hahm HC, Lee CH, Choe JY, Ward A, Lundgren L. Sexual Attitudes, Reasons for Forgoing Condom Use, and the Influence of Gender Power among Asian-American Women: A Qualitative Study. J AIDS Clin Res. 2011 Dec 30;(S1):004. doi: 10.4172/2155-6113.S1-004. PMID 22866240
- [Background] Lee J, Hahm HC. HIV risk, substance use, and suicidal behaviors among Asian American lesbian and bisexual women. AIDS Educ Prev. 2012 Dec;24(6):549-63. doi: 10.1521/aeap.2012.24.6.549. PMID 23206203
- [Background] Hahm HC, Jang J, Vu C, Alexander LM, Driscoll KE, Lundgren L. Drug use and suicidality among Asian American women who are children of immigrants. Subst Use Misuse. 2013 Dec;48(14):1563-76. doi: 10.3109/10826084.2013.808219. Epub 2013 Jul 12. PMID 23848381
- [Background] Hahm HC, Gonyea JG, Chiao C, Koritsanszky LA. Fractured Identity: A Framework for Understanding Young Asian American Women's Self-harm and Suicidal Behaviors. Race Soc Probl. 2014;6(1):56-68. doi: 10.1007/s12552-014-9115-4. PMID 24563680
- [Background] Hahm HC, Chang ST, Tong HQ, Meneses MA, Yuzbasioglu RF, Hien D. Intersection of suicidality and substance abuse among young Asian-American women: implications for developing interventions in young adulthood. Adv Dual Diagn. 2014;7(2):90-104. doi: 10.1108/ADD-03-2014-0012. PMID 25031627
- [Background] Augsberger A, Yeung A, Dougher M, Hahm HC. Factors influencing the underutilization of mental health services among Asian American women with a history of depression and suicide. BMC Health Serv Res. 2015 Dec 8;15:542. doi: 10.1186/s12913-015-1191-7. PMID 26645481
- [Background] Hahm HC, Lee J, Chiao C, Valentine A, Le Cook B. Use of Mental Health Care and Unmet Needs for Health Care Among Lesbian and Bisexual Chinese-, Korean-, and Vietnamese-American Women. Psychiatr Serv. 2016 Dec 1;67(12):1380-1383. doi: 10.1176/appi.ps.201500356. Epub 2016 Jul 1. PMID 27364813

DOCUMENTS (2):
  • Study Protocol (2015-07-24): https://cdn.clinicaltrials.gov/large-docs/49/NCT03370549/Prot_000.pdf
  • Informed Consent Form (2015-08-11): https://cdn.clinicaltrials.gov/large-docs/49/NCT03370549/ICF_001.pdf